CLINICAL TRIAL: NCT05653388
Title: Observational Study of Biomarkers of Disease-related Outcomes in Patients With Metastatic Leiomyosarcoma Receiving Chemotherapy
Brief Title: Metastatic Leiomyosarcoma Biomarker Protocol
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HUM00216516; 1P50CA272170-01 (NIH); HUM00219342 (Other: University of Michigan); HUM00216516 (Other: University of Michigan)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Leiomyosarcoma
Keywords: ctDNA; Biomarker; radiomics
MeSH Terms: conditions — Leiomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional Archival Tissue, Optional Fresh tumor biopsy, blood collections prior to day 1 of first chemotherapy, optional day 8 of cycle 1, day 1 of cycles 2-6 and at progression of sarcoma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Subjects: Once enrolled subjects will provide Optional Archival Tissue, Optional Fresh tumor for a biopsy and blood collections at baseline, optional day 8 of cycle 1, day 1 of cycles 2-6 and at progression
  Interventions: Other: Plasma Collection

INTERVENTIONS:
Other: Plasma Collection — Patients will provide tissue and blood samples. No medical intervention will be completed for study purposes

SUMMARY:
Leiomyosarcoma (LMS) is one of the most prevalent soft tissue sarcomas (STS) and can occur in various sites including soft tissue, uterus and retroperitoneal large vessels. Metastatic disease occurs in approximately 50% of patients diagnosed with leiomyosarcoma and prognosis is poor in setting of metastatic disease. A minority of patients benefit from treatment with chemotherapy and early biomarkers of benefit from treatment are lacking. A biomarker of tumor response and patient survival benefit from chemotherapy early in the course of chemotherapy would be of significant impact in treatment planning. Circulating tumor DNA (ctDNA) is present in blood of patients with advanced/metastatic cancer and may serve as biomarker of tumor response to chemotherapy. Blood samples will be collected prior to and during and chemotherapy, and analyzed for ctDNA and for mutations in genes that are associated with increased risk of developing sarcoma. Tumor tissue will be collected and analyzed for changes in genes. Digital images of the sarcoma from CT or MRI scans obtained during treatment will be obtained for advanced radiomic analysis. Study participants will be asked to complete a questionnaire on attitudes and understanding of genetics and genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic leiomyosarcoma (LMS). There is no age requirement
* Receiving first-line chemotherapy with doxorubicin or gemcitabine/docetaxel
* Target lesions per RECIST 1.1
* Optional archival tumor tissue including 1 H&E-stained slide and unstained tumor tissue [either tissue block containing tumor, or minimum of 4 unstained slides (preferably 8 unstained slides)-fresh frozen sample may also be used in lieu of FFPE sample] available for study research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable or metastatic leiomyosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA with RECIST | 4 years from study start
  To examine the correlation of change in ctDNA with objective tumor response per RECIST. Analysis will occur at each subsequent early time-point (pre-cycle 1 and pre-cycle 2).
Change in ctDNA with progression free survival (PFS) | 54 months from study start
  To examine the correlation of change in ctDNA with progression free survival (PFS). Analysis of ctDNA will occur at each subsequent early time-point (pre-cycle 1 and pre-cycle 2). A Cox regression model will determine whether the baseline ctDNA levels are associated with PFS.

SECONDARY OUTCOMES:
Frequency of ctDNA in patients with unresectable or metastatic leiomyosarcoma. | 4 years from study start
  Plasma collections for ctDNA analysis will be collected at each subsequent early time-point (pre-cycle 1 and pre-cycle 2).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (11):
- United States (9):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Miami, Miami, Florida
  - Dana- Farber, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson, Houston, Texas
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified genetic data on the NIH site, and deidentified imaging data will be shared with the lab at Columbia University. We are not sharing patient identities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the study
Access Criteria: We will share deidentified genetic data on the NIH site, and deidentified imaging data will be shared with the lab at Columbia University. We are not sharing patient identities.